CLINICAL TRIAL: NCT04326088
Title: The Impact of Operation Time and Operators on Postoperative Complication After Free Flap Reconstruction for Patients With Head and Neck Cancer
Brief Title: Postoperative Complication After Free Flap Reconstruction for Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201800440B0
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer; Recurrent Cancer; Surgery--Complications
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- head and neck cancer with free flap reconstruction: patients with head and neck cancer who underwent tumor wide excision and primary free flap reconstruction or secondary free flap reconstruction between March 2008 and February 2017
  Interventions: Other: Reconstruction group; Other: Recurrent group

INTERVENTIONS:
Other: Reconstruction group — Patients with primary tumor which underwent free flap reconstruction group.
Other: Recurrent group — Patients with recurrent tumor which underwent free flap reconstruction group.

SUMMARY:
This study was designed to investigate the outcome of free-flap reconstruction surgery following head and neck cancer resection between primary and recurrent head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck cancer who underwent tumor wide excision and primary free flap reconstruction or secondary free flap reconstruction between March 2008 and February 2017
* Age: 20~100 years old

Exclusion Criteria:

* patients with missing or unvalidated data
* patients less than 20 years old

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2,004 patients with head and neck cancer who underwent tumor wide excision and primary free flap reconstruction or secondary free flap reconstruction between March 2008 and February 2017. After excluding missing or unvalidated data, 1,700 patients with a total of 1,791 free flap reconstructions (21 patients received double free flap reconstructions) was left in the study.
Sampling Method: Probability Sample
Enrollment: 2004 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Failure or success flap | 2 months after surgery
  The condition of the reconstruction flap is failure or success.

SECONDARY OUTCOMES:
Complications | 2 months after surgery
  such as wound infection rate, fistula, hematoma, and partial necrosis of the flap

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No